CLINICAL TRIAL: NCT05975216
Title: Relinking Diagnosed But Untreated HCV Patients Back Into Care.
Acronym: Relink
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Relink
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosed-but-untreated: Diagnosed but untreated (DBU) HCV patients through positive serology with positive or unknown HCV RNA in UZ Brussel between 2012 - 2022.
  Interventions: Other: Contact the patient

INTERVENTIONS:
Other: Contact the patient — Phone call, email or letter to contact the patient to relink them.

SUMMARY:
Reintroduction of patients into a HCV infection care pathway after a positive chronic hepatitis C diagnosis by previous testing in our hospital who were lost in follow-up.

Gaining insight in the possible reasons why patients are lost in follow-up after positive hepatitis C serology.

ELIGIBILITY:
Inclusion Criteria:

* Positive HCV serology between 2012-2022 with positive or uknown HCV RNA in UZ Brussels database
* ≥18 years

Exclusion Criteria:

* Positive HCV serology with negative HCV RNA
* Previously eradicated patients in UZ Brussel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Positive hepatitis C serology with positive or unknown HCV RNA.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Retrospective data collection | before contacting the patient
  Prevalence of diagnosed but untreated HCV patients through positive serology with positive or unknown HCV RNA in UZ Brussel between 2012 - 2022.
Prospective interventional study | from first contact of the patient till 12 weeks after end of treatment.
  To recall DBU patients by phone, e-mail or letter, trying to optimize treated and cured patients after recall

SECONDARY OUTCOMES:
Reason lost in follow-up | from first contact of the patient till 12 weeks after end of treatment.
  Understanding the different reasons why patients were lost in follow-up with the aim of improving our hospital quality in the future:
  * Unaware of positive hep C serology
  * Follow-up or treatment in other centre
  * Refusal of previously proposed therapy
  * Other?

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium